CLINICAL TRIAL: NCT06595446
Title: A Feasibility Randomized Controlled Trial Evaluating Early vs Late Stent Removal Following Radical Cystectomy and Ileal Conduit Formation for Bladder Cancer
Brief Title: A Feasibility Randomized Trial Evaluating Early vs Late Stent Removal Following Radical Cystectomy and Ileal Conduit Formation for Bladder Cancer
Acronym: STENT-OPT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Nicholas Power, Principal Investigator, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 125609
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Bladder Cancer Requiring Cystectomy; Ileal Conduit; Urinary Diversion
Keywords: Bladder cancer; Radical cystectomy; Stent dwell time; Complications; Ileal conduit
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm A (Experimental): Early Stent removal
  Interventions: Procedure: Early Stent removal
- Arm B (Active Comparator): Late Stent removal
  Interventions: Procedure: Late Stent removal

INTERVENTIONS:
Procedure: Early Stent removal — Ureteral JJ stents removed 5-7 days after radical cystectomy and ileal conduit formation
  Arms: Arm A
Procedure: Late Stent removal — Ureteral JJ stents removed 4-6 weeks after radical cystectomy and ileal conduit formation
  Arms: Arm B

SUMMARY:
Bladder cancer is the 4th most common cancer in men and 5th most common type of cancer in Canada. Urothelial cancer accounts for approximately 90% of malignancies. At diagnosis, over 75% of cases are classified as non-muscle invasive (NMIBC), and with appropriate treatment, the majority of these patients achieve positive outcomes. The progression rate of NMIBC to Muscle-invasive bladder cancer (MIBC) varies between 5-50% at 5 years dependent on histopathological features such as grade, stage, presence of CIS and age (Carcinoma in Situ). The optimal treatment of MIBC (T2-T4N0M0) consists of neoadjuvant cisplatin-based chemotherapy followed by Radical cystectomy and urinary diversion (RCUD). In the last couple of decades, RCUD has also gained attention for treating patients with high-risk non-muscle invasive bladder cancer. Despite advancements in surgical techniques and the rise of minimally invasive alternatives, complications after surgery remain frequent, with morbidity rates of approximately 50%.

Several uncertainties persist in surgical practice, including the role of perioperative ureteric stenting during RCUD. Perioperative ureteric stenting is intended to minimize urinary leakage from the newly created uretero-enteric anastomosis and to prevent early obstruction caused by anastomotic swelling. However, stenting may increase the risk of urinary tract infections (UTIs) and necessitate additional follow-up for stent removal. Peng et al. conducted the most recent systematic review in 2021, demonstrating that ureteral stents in RCUD were linked to higher rates of anastomotic strictures. Their review did not provide evidence that these stents were more effective than not using stents in preventing post-diversion urinary leakage. The review underscored the scarcity of prospective randomized controlled trials examining the safety and effectiveness of stenting in this context. The sole prospective (non-randomized) study assessing stent dwell / retention time after RCUD demonstrated early stent removal (2 weeks) had decreased 90-day readmissions and UTIs.

Therefore, the investigators aimed to determine the feasibility of conducting a definitive randomized trial to evaluate patients undergoing radical cystectomy and ileal conduit formation to receive either early stent removal (5-7 days) or late stent removal (4-6 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years or older) undergoing radical cystectomy and ileal conduit formation for bladder cancer
* Able to give informed written consent to participate.

Exclusion Criteria:

* Treatment without curative intent (cT4b, salvage or palliative cystectomies);
* Patients undergoing alternative forms of urinary diversion (e.g. continent cutaneous urinary diversion or orthotopic neobladder formation)
* Patients previously received abdominal/pelvic radiotherapy
* Patients with concomitant upper urinary tract cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Complication rates | within 30 days:
Feasibility Outcomes | 1 year
  1. Recruitment Metrics:
     * Recruitment Rates: Number of participants recruited versus the number of eligible patients.
     * Screen Failures: Number of patients screened but found ineligible.
     * Non-Consenting Rates: Number of eligible patients who decline participation.
  2. Protocol Adherence:
     * Randomization Process Success: Rate of successful randomizations without errors.
     * Protocol Violations / Deviations: Incidents where clinical needs required deviation from the protocol.
     * Completion Rate: Proportion of participants who complete the study according to the protocol.

SECONDARY OUTCOMES:
Complication rates | within 90 days
Readmission rates | within 90 days
Complication rates | within 1 year
  The secondary outcomes will also include composite Uretero-enteric anastomosis (UEA) complications after radical cystectomy and ileal conduit formation.

OTHER OUTCOMES:
Length of stay | 90 days
  Length of inpatient hospital stay following surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Victoria Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beano H, He J, Hensel C, Worrilow W, Townsend W, Gaston K, Clark PE, Riggs S. Safety of decreasing ureteral stent duration following radical cystectomy. World J Urol. 2021 Feb;39(2):473-479. doi: 10.1007/s00345-020-03191-2. Epub 2020 Apr 17. PMID 32303901
- [Background] Peng YL, Ning K, Wu ZS, Li ZY, Deng MH, Xiong LB, Yu CP, Zhang ZL, Liu ZW, Lu HM, Zhou FJ. Ureteral stents cannot decrease the incidence of ureteroileal anastomotic stricture and leakage: A systematic review and meta-analysis. Int J Surg. 2021 Sep;93:106058. doi: 10.1016/j.ijsu.2021.106058. Epub 2021 Aug 18. PMID 34416355
- [Background] Bhindi B, Kool R, Kulkarni GS, Siemens DR, Aprikian AG, Breau RH, Brimo F, Fairey A, French C, Hanna N, Izawa JI, Lacombe L, McPherson V, Rendon RA, Shayegan B, So AI, Zlotta AR, Black PC, Kassouf W. Canadian Urological Association guideline on the management of non-muscle-invasive bladder cancer - Full-text. Can Urol Assoc J. 2021 Aug;15(8):E424-E460. doi: 10.5489/cuaj.7367. No abstract available. PMID 33938798